CLINICAL TRIAL: NCT06275126
Title: Optimizing Surgical Decisions in Young Adults With Breast Cancer
Acronym: CONSYDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-08026433; R01CA256877-01A1 (NIH)
Record Dates: First submitted 2024-02-06; First posted 2024-02-23 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Stage 0; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a pragmatic, Type II hybrid effectiveness-implementation, stepped-wedge design that will incorporate a mixed-methods approach to test the efficacy and evaluate the implementation of the CONSYDER intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Prior to institutional crossover, participants receive care as per usual for 6 months ("run-in" period) and are not sent CONSYDER.
- CONSYDER decision aid (Other): Web-based breast cancer surgery decision aid
  Interventions: Other: CONSYDER decision aid

INTERVENTIONS:
Other: CONSYDER decision aid — Web-based breast cancer surgery decision aid
  Arms: CONSYDER decision aid

SUMMARY:
The goal of this study is to understand and improve the breast surgical decision-making process for young women newly diagnosed with breast cancer. As part of this study, the investigators will evaluate the impact and use a web-based tool called CONSYDER that is designed to provide useful information to young breast cancer patients. It is also meant to improve communication between young women and their surgeons with the purpose of helping patients make appropriate surgical decisions.

Participants will complete surveys approximately within 1 week of the surgical consult and approximately 6 months after surgery. Patients who receive neoadjuvant chemotherapy will also be surveyed after the completion of neoadjuvant treatment but prior to surgery. Some patients will be invited for an interview after their surgery as part of the evaluation. A subset of patients/surgeons will also have their surgical consultation audio-recorded.

DETAILED DESCRIPTION:
Primary objectives:

* To test the effectiveness of the CONSYDER decision support tool on reducing decisional conflict prior to breast cancer surgery.
* To evaluate the implementation of and mechanisms of use for CONSYDER.

Secondary Objectives:

* To determine the impact of CONSYDER on decision-making preferences, breast cancer knowledge, treatment goals and preferences, anxiety, decisional regret, and self-efficacy in communication.

Exploratory Objectives:

* To explore whether CONSYDER impacts surgical choice.

OUTLINE: This is a multi-site cluster randomized trial using a stepped wedge design. Approximately 800 women will be recruited at 4 study sites (Weill Cornell Medicine, Yale Cancer Center, Dana-Farber Cancer Institute, Duke Cancer Institute), including network affiliate sites, over an approximate 30-month period. All sites will have a 6-month "run-in" period where patients will not be sent CONSYDER. The 6-month blocks may be extended if recruitment targets are not met. Sites will be randomized to begin delivery of CONSYDER to all newly diagnosed women, age ≤44, with Stage 0-III breast cancer as part of routine clinical care; young women will have access to the website whether or not they consent to research study participation.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-44
* New diagnosis of Stage 0, 1, 2, or 3 unilateral breast cancer
* English or Spanish speaking

Exclusion Criteria:

* Diagnosis of de novo Stage 4 breast cancer
* Recurrent early-stage breast cancer
* Bilateral breast cancer

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Pre-surgical decisional conflict as measured by the Decisional Conflict Scale (DCS) | pre-surgery
  The Decisional Conflict Scale (DCS) includes 5 subscales (uncertainty, informed, values clarity, support, effective decision). Each item is rated on a scale of 0 (strongly agree)-4 (strongly disagree). Scores range from 0-100 with higher scores indicating more decisional conflict.
Use of CONSYDER pre-consult | pre-surgery
  Proportion of patients eligible to use CONSYDER who logged in prior to surgical consult

SECONDARY OUTCOMES:
Knowledge as measured by adapted Breast Cancer Surgery Decision Quality Instrument (BCS -DQI) | pre-surgery
  Breast cancer knowledge will be assessed using selected questions from the adapted Breast Cancer Surgery Decision Quality Instrument (BCS -DQI), an instrument designed to evaluate the quality of breast cancer treatment decisions. The number of correct responses across (out of a total of 5 items) will be summed.
Treatment goals and preferences as measured by adapted Breast Cancer Surgery Decision Quality Instrument (BCS-DQI) | pre-surgery
  Treatment goals and preferences have been adapted from the BCS-DQI to include preferences salient to young women. We will ask participants to mark on a scale (not important, 0-extremely important, 10) the importance of several reasons in relation to their surgical decision. Ratings for each item will be summarized (e.g., mean, median, range).
Anxiety, as measured with the 8-item Patient Reported Outcomes Measurement Information System (PROMIS) - Anxiety - Short Form | pre-surgery and 6 months post-surgery
  Anxiety, as measured with the 8-item PROMIS - Anxiety - Short Form. Response options for each item range from never (1) to always (5). Raw scores range from 5-40 and T-scores range from 37.1-83.1. Higher scores indicate higher levels of anxiety.
Self-efficacy in communication as measured by the Perceived Efficacy in Patient-Physician Interactions scale (PEPPI). | pre-surgery
  Perceived Efficacy in Patient-Physician Interactions scale (PEPPI) has 5 items. Each item is rated on a (0, not confident at all - 10, extremely confident) scale. Scores range from 0-50, with higher scores indicating greater self-efficacy.
Decisional regret as measured by the Decision Regret Scale (DRS) | 6 months post-surgery
  The Decision Regret Scale (DRS) includes 5 items. Each item is rated on a scale of 1 (strongly agree)-5 (strongly disagree). Scores range from 0-100 (item scores are converted by subtracting "1" from individual items and multiplying by 25). Higher scores indicate more decisional regret.
Receipt of contralateral prophylactic mastectomy | 6 months post-surgery
  Proportion of patients who undergo contralateral prophylactic mastectomy
Fidelity of implementation of CONSYDER via patient portal email | pre-surgical consult
  Proportion of patients eligible to use CONSYDER who were sent an email from patient portal
Use of CONSYDER post-consult | up to 6 months post-surgical consult
  Proportion of patients who logged in to CONSYDER post-surgical consult
Frequency of CONSYDER use pre-consult | pre consult
  Count of the number log-ins to CONSYDER pre-consult
Frequency of CONSYDER use post-consult | up to 6 months post-surgical consult
  Count of the number log-ins to CONSYDER post-consult

CONTACTS AND LOCATIONS:
Overall Officials: Shoshana Rosenberg, ScD, MPH, Principal Investigator — Weill Medical College of Cornell University; Rachel Greenup, MD, MPH, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Yale Cancer Center, New Haven, Connecticut
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medicine, New York, New York
  - Duke Cancer Institute, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sets will made available, by request, to outside researchers. A data use agreement may be required with participating institutions to facilitate sharing of any data sets. Data from qualitative interviews, focus groups, audio-recordings, and any data collected from clinicians/providers will not be made available due to concerns about potentially identifying information being shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available following publication of the primary endpoints of the study. No end date.
Access Criteria: Requests must be made in writing to the principal investigators. A data use agreement may be required with participating institutions to facilitate sharing of any data sets.